CLINICAL TRIAL: NCT02779816
Title: Exploring the Utility of a Novel Adaptive Device for Commercially Available Insulin Pens in Patients With Arthritis or Hand Deformities
Brief Title: Adaptive Device for Insulin Pens for Arthritic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of sufficient recruitment, other priorities
Sponsor: Levenson, David I., M.D. (Individual)
Responsible Party: Principal Investigator, David I. Levenson, MD, PI, Levenson, David I., M.D.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-1
Record Dates: First submitted 2016-05-15; First posted 2016-05-20 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Arthritis
Keywords: Diabetes Mellitus; Arthritis
MeSH Terms: conditions — Diabetes Mellitus; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (pen device) (Experimental): Subjects will use the pen device when using their commercially available insulin pens
  Interventions: Device: Pen device
- Control (No Intervention): Subjects will use the commercially available insulin pens only (no adaptive pen device).

INTERVENTIONS:
Device: Pen device — Adaptive pen device
  Arms: Intervention (pen device)

SUMMARY:
Approximately 34 subjects will be enrolled in an unblinded cross-over design. For one week, they will use the adaptive pen device and for the next week, they will use just the insulin (or other medication) pen. This will be repeated for another one week period each. At the end of each week, the subjects will fill out a questionnaire regarding their experiences and any suggestions for improvements for the design of the pen device.

DETAILED DESCRIPTION:
This study is of an unblinded crossover design. Each patient will be randomly assigned to initiate a one week observation period with either the pen alone or the pen with the device. The following week, the patient will switch to the other assignment. This will be repeated one more time for a total of two weeks with the device and two weeks without it.

At the end of every week, the patients will be given a questionnaire to fill out. Questions will include a measurement of their satisfaction with their insulin (or other medication) delivery system for that week. Patients will be instructed to continue their usual dosage of medication as prescribed by their physician. If the patients have any problems with the device or feel uncomfortable with it, they are instructed to discontinue use of the device and continue using their pen as usual.

The patients may keep the device at the end of the study. The questionnaires that the patients fill out will be the primary source documents.

ELIGIBILITY:
Inclusion Criteria:

* Currently using a pen to administer medication at least once a week
* Currently are having some difficulty (self reported) using their pens because of dexterity issues

Exclusion Criteria:

* Woman of child-bearing age who are known to be pregnant
* People who are unable or unwilling to sign the informed consent document
* Patients who do not understand the proper use of the device after sufficient instruction
* Anyone in the Principal Investigator's judgment who cannot properly use the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for ease of use | one month
  Questionnaires re: efficacy and ease of use

CONTACTS AND LOCATIONS:
Overall Officials: David I Levenson, MD, Principal Investigator — East Coast Medical Associates
Locations (1):
- East Coast Medical Associates, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Not until a patent is approved; after that, upon request